CLINICAL TRIAL: NCT01939223
Title: A Randomized, Double-blind, Placebo-controlled Phase-III Study of Adjuvant Regorafenib Versus Placebo for Patients With Stage IV Colorectal Cancer After Curative Treatment of Liver Metastases
Brief Title: Colorectal Cancer Treated With Adjuvant Regorafenib Versus Placebo After Curative Treatment of Liver Metastases in a Randomized, Double-blind, Placebo-Controlled Phase-III STudy
Acronym: COAST
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15983; 2012-004369-42 (EudraCT Number)
Record Dates: First submitted 2013-09-06; First posted 2013-09-11 (Estimated); Results first posted 2017-10-20 (Actual); Last update posted 2017-10-20 (Actual); Status verified 2017-09

CONDITIONS: Colorectal Neoplasms
Keywords: Stage IV colorectal cancer / Liver Metastasis
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Regorafenib (Experimental): 4 regorafenib tablets taken orally in the morning daily, followed by a low fat meal for 3 weeks on off treatment followed by 1 week off without treatment,Treatment 21 days.
  Interventions: Drug: Regorafenib (Stivarga, BAY73-4506)
- Placebo (Placebo Comparator): 4 placebo tablets taken orally in the morning daily,followed by a low fat meal for 3 weeks on off treatment followed by 1 week off without treatment,Treatment 21 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Regorafenib (Stivarga, BAY73-4506) — Four tablets of 40mg taken orally daily in the morning, dose of 160 mg for 21 days of treatment followed by 7 days without treatment
  Arms: Regorafenib
Drug: Placebo — Four tablets taken in the morning orally daily for 21 days of treatment followed by 7 days without treatment
  Arms: Placebo

SUMMARY:
To evaluate and compare the efficacy and safety of regorafenib versus placebo in subjects with colorectal cancer (CRC) after curative resection of liver metastasis and completion of all planned chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Have a history of a primary adenocarcinoma of the colon and / or rectum
* Have a history of Stage IV Colorectal Cancer (CRC) with metastases to the liver only
* Have received at least 3 months ,of neoadjuvant, adjuvant, or perioperative chemotherapy, including a fluoropyrimidine and either oxaliplatin or irinotecan or both for subjects with initial Stage IV CRC which were treated with surgery with curative intent for both primary and metastatic lesions. The total chemotherapy administered, including that administered prior to and after liver resection, should not exceed 9 months. OR Have received surgery with curative intent for primary CRC and at least 3 months ,of neoadjuvant, adjuvant, or perioperative chemotherapy for the primary tumor, including a fluoropyrimidine or a fluoropyrimidine and either oxaliplatin or irinotecan or both

  * For subjects with liver metastases developing > 6 months after completing treatment for primary CRC and having undergone surgery with curative intent for liver metastases, a second course of chemotherapy lasting at least 3 months needs to be administered, including a fluoropyrimidine and either oxaliplatin or irinotecan or both. The second course of chemotherapy should not exceed 9 months.
* For subjects who developed liver metastases >/=6 months after completing treatment for primary CRC and having undergone surgery with curative intent for liver metastases, a second course of chemotherapy is not permitted unless initial adjuvant therapy consisted of fluoropyrimidine monotherapy. Subjects who received fluoropyrimidine alone must have received a second course of chemotherapy with fluoropyrimidine and either oxaliplatin or irinotecan or both, which should not exceed 9 months.For subjects with initial Stage I or II disease, no chemotherapy is required for a primary CRC lesion treated with surgery with curative intent. These subjects must receive chemotherapy for the treatment of liver metastases (which were also treated with surgery with curative intent), which must last at least 3 months, including a fluoropyrimidine and either oxaliplatin or irinotecan or both. The total course of chemotherapy should not exceed 9 months.
* Prior to randomization, have histological confirmation that CRC lesions were adenocarcinoma (subtypes of adenocarcinoma, e.g. mucinous adenocarcinoma are allowed). Subjects with CRC lesions of other histological types, including mixed type with predominant adenocarcinoma, will not be eligible to be randomized to study treatment.
* Have pathology-proven complete removal of all primary and liver metastatic CRC lesions. Subjects with positive margins will not be eligible for the study.
* Have adequate bone marrow function, liver function, and renal function, as measured by the following laboratory assessments conducted within 7 days prior to the initiation of study treatment:

  * Total bilirubin </=1.5 times the upper limit of normal (ULN)
  * Alanine aminotransferase and aspartate aminotransferase </= 3 times the ULN
  * Lipase</=1.5 times the ULN
  * Serum creatinine</=1.5 times the ULN
  * Carcinoembryonic antigen (CEA)</=3 times the ULN
  * Glomerular filtration rate>/=30 mL/min/1.73 m2 according to the Modified Diet in Renal Disease abbreviated formula
  * International normalized ratio of prothrombin time and activated partial thromboplastic time </=1.5 times the ULN. Subjects who are therapeutically treated with an agent such as warfarin or heparin will be allowed to participate if no underlying abnormality in coagulation parameters exists per medical history.
  * Platelet count >/=100,000 /mm3, hemoglobin >/=9 g/dL, absolute neutrophil count >/= 1500/mm3 without transfusions or granulocyte colony stimulating factor and other hematopoietic growth factors
  * Alkaline phosphatase ≤ 2.5 times the ULN
* Have had a CT or MRI scan (chest, abdomen, pelvis and other suspected sites as applicable) to determine eligibility for randomization within 4 weeks prior to randomization (hereafter referred to as the "eligibility scan")
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 14 days prior to the initiation of study treatment
* If female and of childbearing potential, or if male, agree to use adequate contraception (e.g., abstinence, intrauterine device, oral contraceptive, or double barrier method) based on the judgment of the investigator or a designated associate from the date on which the ICF is signed until 8 weeks after the last dose of study drug.

Exclusion Criteria:

* Are taking strong cytochrome P (CYP) CYP3A4 inhibitors (eg, clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, posaconazole, ritonavir, saquinavir, telithromycin, voriconazole) or strong CYP3A4 inducers (eg, carbamazepine, phenobarbital, phenytoin, rifampin, St. John's Wort).
* Have used biologic response modifiers, such as granulocyte-colony stimulating factor, within 3 weeks prior to signing the ICF.
* Have had prior treatment with regorafenib or any other (vascular endothelial growth factor receptor) VEGFR-targeting kinase inhibitor.
* Have had anti-cancer treatment following liver resection that exceeded a duration of 6 months.
* Have been treated with biologics (eg, antibodies targeting VEGFR or EGFR) after liver resection unless the administration of the biologic started prior to liver resection and continued after liver resection only to complete a pre-specified number of cycles.
* Completed their last dose of chemotherapy or had their last cancer surgery more than 10 weeks, whichever came later, prior to randomization.
* Have extra-hepatic metastatic disease. Suspicious lesions should be rigorously evaluated with other imaging techniques and/or biopsy to exclude extra-hepatic metastatic disease prior to submitting for central radiology review.
* Have had systemic anticancer therapy including cytotoxic therapy, signal transduction inhibitors, immunotherapy, and/or hormonal therapy within 4 weeks prior to initiation of study treatment.
* Are pregnant and or breast feeding.
* Have had prior or concurrent cancer distinct in primary site or histology from CRC within 5 years prior to randomization EXCEPT for curatively treated cervical cancer in situ, nonmelanoma skin cancer, Stage 0 intramucosal gastric cancer after endoscopic complete removal, or superficial bladder tumors classified as noninvasive tumor (Ta), carcinoma in situ (Tis), or tumor invades lamina propria (T1).
* Have congestive heart failure classified as New York Heart Association Class 2 or higher.Have had unstable angina (angina symptoms at rest) or new-onset angina ≤ 3 months prior to screening. Have had a myocardial infarction < 6 months prior to initiation of study treatment.
* Have cardiac arrhythmias requiring anti-arrhythmic therapy, with the exception of beta blockers or digoxin.
* Have uncontrolled hypertension (systolic blood pressure [SBP] greater than140 mmHg or diastolic blood pressure [DBP] greater than 90 mmHg) despite optimal medical management.
* Have pheochromocytoma.
* Have had arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis, or pulmonary embolism within 6 months prior to the initiation of study treatment.
* Have a known history of human immunodeficiency virus infection.
* Have either active or chronic hepatitis B or C requiring treatment with antiviral therapy.
* Have a seizure disorder requiring medication.
* Have evidence or history of any bleeding diathesis (including mild hemophilia), irrespective of severity.
* Have had a hemorrhage or a bleeding event >/=Grade 3 (NCI-CTCAE v 4.0) within 4 weeks prior to the initiation of study treatment.
* Have any other serious or unstable illness, or medical, social, or psychological condition, that could jeopardize the safety of the subject and/or his/her compliance with study procedures, or may interfere with the subject's participation in the study or evaluation of the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-12-02 (Actual); Primary Completion 2016-08-29 (Actual); Study Completion 2016-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (100):
- United States (20):
  - Laguna Hills, California
  - Los Angeles, California
  - New Haven, Connecticut
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Detroit, Michigan
  - Rochester, Minnesota
  - Omaha, Nebraska
  - New Brunswick, New Jersey
  - Buffalo, New York
  - New York, New York
  - Syracuse, New York
  - Duke University Medical Center, Durham, North Carolina
  - Philadelphia, Pennsylvania
  - Chattanooga, Tennessee
  - Germantown, Tennessee
  - Dallas, Texas
  - Richmond, Virginia
  - Kirkland, Washington
  - Seattle, Washington
- Australia (4):
  - Liverpool, New South Wales
  - East Melbourne, Victoria
  - Bentleigh East
  - Malvern
- Belgium (3):
  - Edegem
  - Leuven
  - Liège
- Brazil (4):
  - Belo Horizonte, Minas Gerais
  - Porto Alegre, Rio Grande do Sul
  - São José do Rio Preto, São Paulo
  - São Paulo, São Paulo
- Canada (4):
  - Edmonton, Alberta
  - Toronto, Ontario
  - Sherbrooke, Quebec
  - Montreal
- China (10):
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Guangzhou, Guangdong
  - Harbin, Heilongjiang
  - Wuhan, Hubei
  - Changsha, Hunan
  - Xi'an, Shaanxi
  - Kunming, Yunnan
  - Hangzhou, Zhejiang
  - Beijing
  - Shanghai
- France (9):
  - Bordeaux
  - Brest
  - Clermont-Ferrand
  - Lyon
  - Marseille
  - Paris
  - Poitiers
  - Tours
  - Villejuif
- Germany (5):
  - München, Bavaria
  - Frankfurt am Main, Hesse
  - Oldenburg, Lower Saxony
  - Mainz, Rhineland-Palatinate
  - Berlin
- Israel (3):
  - Haifa
  - Ramat Gan
  - Tel Aviv
- Italy (9):
  - Foggia, Apulia
  - Napoli, Campania
  - Reggio Emilia, Emilia-Romagna
  - Udine, Friuli Venezia Giulia
  - Rome, Lazio
  - Brescia, Lombardy
  - Milan, Lombardy
  - Florence, Tuscany
  - Pisa, Tuscany
- Japan (17):
  - Kashiwa, Chiba
  - Sapporo, Hokkaido
  - Akashi, Hyōgo
  - Amagasaki, Hyōgo
  - Kobe, Hyōgo
  - Kasama, Ibaraki
  - Yokohama, Kanagawa
  - Suita, Osaka
  - Takatsuki, Osaka
  - Sunto, Shizuoka
  - Shimotsuke, Tochigi
  - Koto-ku, Tokyo
  - Minato-ku, Tokyo
  - Mitaka, Tokyo
  - Shinagawa, Tokyo
  - Shinjuku-ku, Tokyo
  - Fukuoka
- Portugal (3):
  - Almada
  - Porto
  - Santa Maria da Feira
- Spain (6):
  - Alicante
  - Badajoz
  - Barcelona
  - Córdoba
  - Madrid
  - Valencia
- United Kingdom (3):
  - Royal Marsden NHS Trust (Surrey), Sutton, Surrey
  - Bristol
  - London

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multinational study was conducted at 32 study centers that screened 65 subjects across 9 countries, between 02 December 2013 (start of enrollment) and 29 August 2016 (last patient last vist).
Pre-assignment Details: Overall, 65 subjects were screened, of which 40 were screen failures. The remaining 25 subjects were randomized and assigned to treatment. All 25 subjects received treatment.
Groups:
- Regorafenib 160 mg: Description: Subjects received regorafenib 160 milligram (mg) (4 * 40 mg tablets) orally once daily on a 3 weeks on / 1 week off dosing schedule.
- Placebo: Subjects received placebo matching to regorafenib tablet orally once daily on a 3 weeks on / 1 week off dosing schedule.
Period: Overall Study
Arm/Group | Regorafenib 160 mg | Placebo
Started | 14 | 11
Participants Received Treatment | 14 | 11
Completed | 1 | 0
Not Completed | 13 | 11
Not completed — AE not assoc. with disease recurrence | 1 | 1
Not completed — Disease recurrence (radiological) | 1 | 3
Not completed — Study stopped by Sponsor | 5 | 7
Not completed — Withdrawal by Subject | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Regorafenib 160 mg | Placebo | Total
Number analyzed (Participants) | 14 | 11 | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.7 (11.22) | 57.0 (9.83) | 58.5 (10.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Disease Free Survival (DFS) as Assessed by the Investigator
Description: Disease free survival was evaluated by CT / MRI scans as assessed by the investigator, which was defined as the time (in days) from date of randomization to date of first observed radiographic disease recurrence (RECIST 1.1 criteria for measurable and non-measurable disease) or death due to any cause, if death occurred before disease recurrence was documented. For subjects without documented disease recurrence or death at the time of analysis, the DFS time was censored at the date of the last evaluable CT / MRI scan.
Time Frame: From date of randomization to date of first observed radiographic disease recurrence (RECIST 1.1 criteria for measurable and non-measurable disease) or death due to any cause, if death occurred before disease recurrence was documented.
Population: Number of Participants Analyzed is 0 because this study was prematurely terminated and data were not collected for this endpoint.
Arm/Group | Regorafenib 160 mg | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as the time (days) from randomization to death due to any cause. The OS time for subjects alive at the time of analysis was censored at their last date known to be alive.
Time Frame: Subjects who experienced disease recurrence (either during treatment or during Active Follow-up), or otherwise withdrew from the study for any reason other than death, were followed for overall survival unless consent was withdrawn.
Population: as for outcome 1
Arm/Group | Regorafenib 160 mg | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From the start of study drug administration until 30 days after the last study medication intake.
Groups:
- Regorafenib 160 mg (BAY73-4506): Subjects received regorafenib 160 mg (4 *40 mg tablets) orally every day for 3 weeks followed by 1 week off treatment plus BSC (best supportive care).
- Placebo: Subjects received placebo matched to regorafenib tablets orally every day for 3 weeks followed by 1 week off treatment plus BSC (best supportive care).
Arm/Group | Regorafenib 160 mg (BAY73-4506) | Placebo
Serious Adverse Events (participants affected / at risk) | 2/14 | 0/11
Other Adverse Events (participants affected / at risk) | 13/14 | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regorafenib 160 mg (BAY73-4506) (N=14) | Placebo (N=11)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Generalised erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regorafenib 160 mg (BAY73-4506) (N=14) | Placebo (N=11)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abscess oral (Infections and infestations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (6) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 2 (4) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 4 (10) | 0 (0)
Asthenia (General disorders) | 4 (6) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 5 (7) | 0 (0)
Blood bilirubin unconjugated increased (Investigations) | 1 (2) | 0 (0)
Blood creatinine decreased (Investigations) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 3 (3) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (5) | 2 (2)
Contrast media allergy (Immune system disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (5)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (2) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Fatigue (General disorders) | 2 (2) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (2) | 1 (1)
Generalised erythema (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Genital infection fungal (Infections and infestations) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Glycosuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Hair follicle tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (2) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (4) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 7 (29) | 1 (2)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 4 (7) | 1 (4)
Lymphocyte count decreased (Investigations) | 1 (2) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (2)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (3) | 0 (0)
Neutrophil count increased (Investigations) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 6 (22) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (3) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 4 (9) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Pyrexia (General disorders) | 3 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rhinitis atrophic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (3) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (4) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Weight increased (Investigations) | 0 (0) | 1 (2)
White blood cell count decreased (Investigations) | 3 (5) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0)
White blood cells urine positive (Investigations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was prematurely terminated. Analysis was not performed for primary and secondary outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other